CLINICAL TRIAL: NCT04395703
Title: Barriers, Challenges and Facilitators for the Unicef Baby Friendly Initiative (BFI): A Qualitative Study of Maternity Staff Experiences
Brief Title: Baby Friendly Initiative Implementation: Maternity Staff Experiences
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Dorset County Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 274438
Record Dates: First submitted 2020-05-12; First posted 2020-05-20 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Experience, Life
Keywords: Staff experience,barriers,challenges,facilitators
MeSH Terms: interventions — Interviews as Topic; Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maternity staff: Interviews with maternity staff working within a maternity unit including midwifery managers and infant feeding lead staff members.
  Interventions: Other: Interviews and focus groups
- Neonatal unit staff: Staff working within a local maternity unit.
  Interventions: Other: Interviews and focus groups

INTERVENTIONS:
Other: Interviews and focus groups — Unstructured and semi-structured interviews with open ended questions.

SUMMARY:
This qualitative, case study will explore the experiences of maternity staff in England when implementing the World Health Organisation and Unicef Baby Friendly Initiative (BFI) standards within a maternity organisation.

DETAILED DESCRIPTION:
A range of maternity staff over 4 UK NHS hospitals will be recruited and interviewed by one chief investigator regarding their experiences of working with the BFI standards in their daily professional practice.

ELIGIBILITY:
Inclusion criteria

* Maternity staff who have had training in and with experience of working with the BFI.
* Senior neonatal staff working in the maternity unit.
* Maternity unit management.
* Staff in specialised infant feeding roles at local hospitals.
* Student midwives on placement at main study hospital site.
* English speaking.

Exclusion criteria

* Maternity staff with no BFI experience.
* Medical staff.
* Community maternity staff.
* Community nurses and health visitors.
* Student nurses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maternity and neonatal staff who meet the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
To identify barriers to the successful implementation of Unicef Baby Friendly Initiative within a maternity organisation. | 2 years
  The aim is to identify themes regarding barriers that are in place when implementing policies into maternity organisations. These will be developed into recommendations which managers and policy makers can utilise to enable change management.
To identify challenges to the successful implementation of Unicef Baby Friendly Initiative within a maternity organisation. | 2 years
  The aim is to identify themes regarding the challenges that are in place when implementing policies into maternity organisations. These will be developed into recommendations which managers and policy makers can utilise to enable change management.
To identify what facilitates the successful implementation of Unicef Baby Friendly Initiative within a maternity organisation. | 2 years
  The aim is to identify themes regarding the facilitators when implementing the Unicef Baby Friendly Initiative into maternity organisations. These will be developed into recommendations which managers and policy makers can utilise to enable change management.

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Tennant, Principal Investigator — Postgraduate Researcher and Midwife
Locations (1):
- Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: No